CLINICAL TRIAL: NCT02316041
Title: Clinical Trial of the Femtosecond Laser System VisuMax for Refractive Correction of Hyperopia by Means of Lenticule Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tilganga Institute of Ophthalmology (Other)
Collaborators: London Vision Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177/2013
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Hyperopia
Keywords: Femtosecond laser; Small incision lenticule extraction (SMILE)
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Small incision lenticule extraction (Experimental): Small incision lenticule extraction (SMILE) is a form of corneal laser refractive surgery performed using a femtosecond laser
  Interventions: Procedure: Small incision lenticule extraction; Device: ReLEx® (SMILE)

INTERVENTIONS:
Procedure: Small incision lenticule extraction — The VisuMax femtosecond laser is used to create two interfaces that define a refractive lenticule of stromal tissue and a 2mm wide tunnel to connect the upper layer to the corneal surface. The lenticule is manually dissected and removed through the small 2mm incision without the need to create a flap as in LASIK.
  Other Names: SMILE; Refractive lenticule extraction; ReLEx
Device: ReLEx® (SMILE)

SUMMARY:
This is a feasibility and clinical evaluation study of the VisuMax femtosecond laser for refractive correction of hyperopia using the small incision lenticule extraction (ReLEx smile) method.

In ReLEx® the VisuMax femtosecond laser creates two interfaces that define a refractive lenticule of stromal tissue. In ReLEx® FLEx, the upper interface is converted into a LASIK flap by the creation of a sidecut. The LASIK flap is lifted and the lenticule can be removed to correct the refractive error by tissue subtraction. In ReLEx® smile, the lenticule is dissected and removed through a small 2-3mm incision without the need to create a whole flap.

The aims are i) to optimize the VisuMax settings for lenticule separation ii) to optimize the lenticule geometry iii) to assess the safety, efficacy and stability of the treatment

ELIGIBILITY:
Inclusion Criteria:

* older than 21 years of age,
* maximum hyperopic meridian between +1.00D and +7.00D
* astigmatism up to 6D
* CDVA of:

  1. 20/200 or worse in the eye(s) being treated for Phase I
  2. Between 20/200 and 20/100 in the eye(s) being treated for Phase II
  3. Between 20/40 and 20/60 in the eye(s) being treated for Phase III
  4. 20/25 or better for Phase IV
* total uncut stromal thickness of more than 300 µm
* no previous refractive surgery,
* no ocular disease,
* normal corneal topography,
* contact lens wearers have to stop wearing hard contact lenses at least 4 weeks and soft contact lenses 2 weeks prior to pre-examination,
* willing to attend follow-up examinations within the scope of the clinical investigation,
* able and willing to sign the informed consent

Exclusion Criteria:

* patients who are not being able to lie flat in a horizontal position,
* patients who are not being able to understand and give informed consent,
* pregnant or nursing women (or women who are planning to became pregnant during the clinical investigation),
* diagnosis of an autoimmune disease (e.g. AIDS), connective tissue disease or diabetes,
* treatment with medications such as steroids or immune-suppressants,
* herpes simplex or herpes zoster keratitis,
* all standard medical exclusion criteria for LASIK

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety of corrected distance visual acuity (change in corrected distance visual acuity) | 1 year
  Assess the change in corrected distance visual acuity (CDVA) before and after the SMILE procedure.
Efficacy of uncorrected distance visual acuity (uncorrected distance visual acuity achieved after the SMILE procedure relative to the preoperative CDVA) | 1 year
  Measure the uncorrected distance visual acuity achieved after the SMILE procedure relative to the preoperative CDVA for all eyes where the intended target refraction was emmetropia.
Predictability of refractive outcome ( change in manifest refractive error) | 1 year
  Measure the change in manifest refractive error (sphere, cylinder, spherical equivalent) after the SMILE procedure and analyze the predictability relative to the intended target refraction as well as the refractive stability over the 1 year follow-up period

SECONDARY OUTCOMES:
Optical zone centration (Measure the achieved centration of the optical zone) | 1 year
  Measure the achieved centration of the optical zone by topography relative to the corneal vertex (the intended treatment center)
Optical zone diameter | 1 year
  Measure the achieved optical zone diameter from tangential curvature difference maps relative to the intended optical zone

CONTACTS AND LOCATIONS:
Overall Officials: Kishore R Pradhan, MD, Principal Investigator — Tilganga Institute of Ophthalmology
Locations (1):
- Tilganga Institute of Ophthalmology, Refractive Surgery Unit, Kathmandu, Nepal

REFERENCES:
- [Background] Blum M, Kunert KS, Vossmerbaumer U, Sekundo W. Femtosecond lenticule extraction (ReLEx) for correction of hyperopia - first results. Graefes Arch Clin Exp Ophthalmol. 2013 Jan;251(1):349-55. doi: 10.1007/s00417-012-2064-y. Epub 2012 Jun 14. PMID 22695934